CLINICAL TRIAL: NCT06772974
Title: Comparison of Tablet Ginger Versus Tablet Doxylamine Succinate in Control of Nausea and Vomiting in Pregnancy
Brief Title: Tablet Ginger Versus Tablet Doxylamine Succinate in Control of Nausea and Vomiting in Pregnancy
Acronym: GDNVP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nawaz Sharif Medical College (Other)
Collaborators: University of Gujrat (Other)
Responsible Party: Principal Investigator, Zunaira Pervez, Post Gradute Resident, Nawaz Sharif Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GingerVsDoxylamine; NSMC/GYNOBS/14/25 (Other: Nawaz Sharif Medical College); NCT06772974 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Nausea Gravidarum; Hyperemesis Gravidarum
Keywords: Nausea; Vomiting; Pregnancy
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginger Group (Experimental): Ginger
  Interventions: Dietary Supplement: Ginger
- Doxylamine Group (Active Comparator): Tab. Doxylamine Succinate USP
  Interventions: Drug: Doxylamine Succinate USP

INTERVENTIONS:
Drug: Doxylamine Succinate USP — Tab. Doxylamine Succinate
  Arms: Doxylamine Group
Dietary Supplement: Ginger — Ginger (zingiber officinale)
  Arms: Ginger Group

SUMMARY:
Nausea and vomiting are common GI symptoms of pregnancy. Multiple managing options have been used for NVP. Doxylamine succinate is used as first line treatment for NVP despite that alternative modalities such as ginger extracts and tablets is being explored.

This RCT will be conducted after taking ethical approval and informed consent, in Department of Gynecology, Aziz Bhatti Shaheed teaching hospital, Gujrat. Patients will be divided into two equal groups. One group will receive tablet ginger while other group will receive Doxylamine succinate tablets. Baseline PUQE score (3- 15 point scale) over 24 hour will be noted according to symptoms of nausea and vomiting following 7 days of treatment and then at 2nd and 3rd week. Comparison of the change in the severity of nausea from baseline scores (Post-therapy PUQE score - base line scores) in both groups will be considered for results.

DETAILED DESCRIPTION:
Nausea and vomiting are the most common gastrointestinal symptoms of pregnancy. Several treatments have been used for managing NVP. Multiple medications have been used in treatment of NVP. Doxylamine plus pyridoxine is used as first line therapy for NVP. However treatment with alternative medications including ginger extracts and tablets is being explored.

This randomized control trial will be conducted after taking ethical approval and informed consent, in Department of Gynecology, Aziz Bhatti Shaheed teaching hospital, Gujrat. Total 66pregnant females will be enrolled. Demographical data will be recorded. Patients will be divided into two groups (n= 33 in each group). Group A will receive tablet ginger (Zingiber officinale 250mg orally four times daily for 21 days). Group B will receive Doxylamine succinate tablets (10 mg orally, three times daily for 21 days). Baseline PUQE score (3- 15 point scale) over 24 hour will be noted according to symptoms of nausea and vomiting following 7 days of treatment and then at 2nd and 3rd week. Comparison of the change in the severity of nausea from baseline scores (Post-therapy PUQE score - base line scores) in both groups.

Data will be analyzed via SPSS version 25.0. Independent t test and Chi-square test will be used for comparison of the variables between the groups. A paired t test will be used to assess the mean difference in PUQE score within each group (baseline to follow-up). A p-value ≤ 0.05 will be considered as significant. This study aims to compare the efficacy of these two interventions in controlling or reducing the NVP in pregnant women particularly in our local population and will also explore whether ginger or Doxylamine succinate is better in terms of safety. The study will have both theoretical and practical implications provides evidence based clinical data regarding effective NVP treatment in our local population. However, the study will be limited to single center and small sample size.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age>18 years
* 5 to 8weeks of gestation and 8+1to11weeks
* Attending OPD with signs and symptoms of nausea and vomiting with ultrasound confirmed pregnancy
* 1st and 2nd gravida
* Patients who will give consent

Exclusion Criteria:

* Patients were hospitalized for Hyperemesis Gravidarum
* Medical disorders like Diabetes Mellitus, Hepatic, Gastric, Pancreatic, Pyelonephritis, Thyroid and Psychological Disorder
* Patients not responding to treatment after 1week will be excluded
* Patients who will not give consent

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in Nausea and Vomiting based on Pregnancy-Unique Quantification of Emesis Score | 21 Days
  improvement in Nausea and reduction in Vomiting based on Pregnancy-Unique Quantification of Emesis score. This score depicts the severity of emesis. Mild 4-6 moderate 7-12 and severe emesis is considered when score is more than 13. The primary efficacy endpoint will be the change from baseline in PUQE score after 21 days (± 1 day).

SECONDARY OUTCOMES:
Side Effects of Treatment | 21 Days
  The secondary outcomes will include the adverse effects like headache, sedation, constipation, heart burning or any other effect that will be reported by patient.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Shaista Waheed Professor, MBBS, FCPS, Study Director — Nawaz Sharif Medical College, Gujrat
Locations (1):
- Aziz Bhatti Shaheed Teaching Hospital, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Privacy of patients

REFERENCES:
- [Background] Hu Y, Amoah AN, Zhang H, Fu R, Qiu Y, Cao Y, Sun Y, Chen H, Liu Y, Lyu Q. Effect of ginger in the treatment of nausea and vomiting compared with vitamin B6 and placebo during pregnancy: a meta-analysis. J Matern Fetal Neonatal Med. 2022 Jan;35(1):187-196. doi: 10.1080/14767058.2020.1712714. Epub 2020 Jan 14. PMID 31937153